CLINICAL TRIAL: NCT03734445
Title: Effect of Vitamin C, Vitamin D and Zinc Supplementation on the Immune and Inflammatory Process in Type 2 Diabetic Subjects in Mexico
Brief Title: Effect of Vitamin C, D and Zinc Supplementation on the Immune and Inflammatory Process in Type 2 Diabetic Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma del Estado de Mexico (Other)
Responsible Party: Principal Investigator, Roxana Valdés Ramos, DSc, Head of Nutrition and Health Group, Full-time professor, Universidad Autonoma del Estado de Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/11
Record Dates: First submitted 2018-07-05; First posted 2018-11-08 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus type 2; Vitamin C; Vitamin D; Cinc
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly allocated to two groups (vitamin supplement or placebo), with a duration of 24 weeks. Dietary and compliance monthly follow-up and baseline, 12 and 24-week measurements.
Who Masked: Participant, Investigator
Masking Description: Vitamin Supplement and placebo will be packaged by others not including the investigators, code will be kept secret until the end of the trial or unless a secondary effect is registered and merits the opening of the code
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin supplement (Experimental): Effervescent tablets containing Vitamin C, Vitamin D and zinc
  Interventions: Dietary Supplement: Vitamin Supplement
- Placebo (Placebo Comparator): Effervescent tablets not containing Vitamin C, Vitamin D and zinc
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin Supplement — Subjects will be randomly allocated to a supplementation of vitamin C 1000mg, vitamin D 400 IU and zinc 10 mg or an identical placebo. Subjects and researchers will be blinded to the supplement or placebo in order to guarantee double-blinding
  Arms: Vitamin supplement
Other: Placebo — Subjects will be randomly allocated to a supplementation of an identical placebo. Subjects and researchers will be blinded to the supplement or placebo in order to guarantee double-blinding
  Arms: Placebo

SUMMARY:
Type 2 Diabetes Mellitus According to the World Health Organization (WHO), there are more than 346 million individuals with diabetes, of which 90% are type 2. Global estimations for the year 2030 predict an epidemic increase that will reach 366 million. According to the National Nutrition and Health Survey of 2006 (ENSANUT2005), there are 6.4 million type 2 diabetic subjects in Mexico.

According to the calculation of the sample size, the investigators will include 120 adults with type 2 diabetes mellitus selected from the outpatient preventive medicine offices of health centres in the State of Mexico who will divided in two groups: supplement and placebo (60 per group). After having been invited to participate and obtaining the informed consent, study subjects will be evaluated for dietary information, as well as biochemical biomarkers of metabolic control, anthropometric, immune and inflammatory markers, gut microbiota and oxidative stress, before beginning the trial, and after 12 and 24 weeks of supplementation. They will have a monthly follow-up visit for evaluation of adherence and adverse effects, as well as delivery of the supplement.

DETAILED DESCRIPTION:
Subjects will be randomly allocated to a supplementation with 1000 mg vitamin C, 400 IU vitamin D and 10 mg of zinc or placebo group, during 24 weeks. Subjects and researchers will be blinded to the supplement or placebo in order to guarantee double-blinding.

ELIGIBILITY:
Inclusion Criteria:

* Between 25 and 55 years of age, as this is the age in which type 2 diabetes mellitus is more prevalent and there is less probability of encountering multiple diseases in the same subjects
* Both sexes
* Outpatients
* BMI ≥ 25

Exclusion Criteria:

* Without any other chronic disease (cancer, cardiovascular diseases, arthritis and Alzheimer's).
* Severe renal insufficiency.
* Nephrolithiasis or history of nephrolithiasis.
* Hyperoxaluria.
* Hemochromatosis.
* Hypercalcaemia.
* Hypervitaminosis D.
* Using insulin.
* Be taking drugs such as desferrioxamine, iron, cyclosporine, indinavir (protease inhibitors), warfarin, thiazide diuretic, orlistat, ion exchange resins (e.g cholestyramine, laxatives (e.g. mineral oil, senna), vitamin d analogues (e.g. ergocalciferol, calcitriol, and topical calcipotriene), tetracycline antibiotics, quinolone antibiotics, penicillamine, biphosphonates, levothyroxine, eltrombopag.
* Patients with hypersensitivity to any of the active substance(s) or to any of the excipients.
* Hypersensitivity to the by-products including honey, conifers, poplars, Peru balsam, and salicylate.
* Intake of probiotics or supplemental vitamin or mineral (vitamin D, C, zinc or calcium) for 4 weeks before the beginning of the study.
* Smoking and alcohol consumption (> 40 gr/ day for men and 25 gr/ day for women.
* Pregnant or lactating.
* Whose parents or grandparents are/were immigrant or of native origin.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-09 (Estimated); Primary Completion 2020-01-09 (Estimated); Study Completion 2020-03-26 (Estimated)

PRIMARY OUTCOMES:
Change in glycemia from baseline to 12 and 24 weeks | Baseline, 12 and 24 weeks
  Measured in plasma with a Selectra II automated equipment with Randox reactants, in mg/dL
Change in glycosilated Hemoglobin (Hb1Ac) from baseline to 12 and 24 weeks | Baseline, 12 and 24 weeks
  Measured in plasma with a Selectra II automated equipment with Randox reactants, in percentage
Change in plasma insulin from baseline to 12 and 24 weeks | Baseline, 12 and 24 weeks
  Multiplex Technology in a Milliplex Luminex Equipment with Merck-Millipore reactants, in uU/mL
Change in Homeostatic Model Assesment for Insulin Resistance (HOMA-IR) from baseline to 12 and 24 weeks | Baseline, 12 and 24 weeks
  Calculated from: HOMA-IR = (insulin x glucose)/405

SECONDARY OUTCOMES:
Change in plasma cytokines from baseline to 12 and 24 weeks | Baseline, 12 and 24 weeks
  Tumor Necrosis Factor alfa (TNFα), Interferon gamma (IFN-γ), Interleukins 1 beta, 4, 6 and 10 (IL-1β, IL4, IL-6, IL10) & transforming growth factor beta (TGF-β), measured with Multiplex Technology in a Milliplex Luminex Equipment with Merck-Millipore reactants, in pg/mL
Change in plasma adipokines from baseline to 12 and 24 weeks | Baseline, 12 and 24 weeks
  Adiponectin, resistin and leptin, measured with Multiplex Technology in a Milliplex Luminex Equipment with Merck-Millipore reactants, in pg/mL
Change in additional plasma inflammatory markers from baseline to 12 and 24 weeks | Baseline, 12 and 24 weeks
  Apolipoproteins A and B, C-reactive protein, vascular cell adhesion protein (V-CAM), intercellular adhesion molecule (I-CAM), complement proteins C-3 and C-4, measured with Multiplex Technology in a Milliplex Luminex Equipment with Merck-Millipore reactants, in pg/mL
Change in lipid profile from baseline to 12 and 24 weeks | Baseline, 12 and 24 weeks
  Total cholesterol, HDL-, LDL-, Very Low Density Lipoprotein (VLDL)-cholesterol and triacylglycerides, measured in plasma with a Selectra II automated equipment with Randox reactants, in mg/dL
Changes in markers of oxidative stress from baseline to 12 and 24 weeks | Baseline, 12 and 24 weeks
  Malondialdehyde (QuantiChromTM), Thiobarbituric acid reactive substances (TBARS Assay Kit), carbonylated proteins (colorimetric), antioxidant capacity (QuantiChromTM Antioxidant Assay Kit), catalase (EnzyChromTM Catalase Assay Kit), superoxide dismutase (EnzyChromTM Superoxide Dismutase Assay Kit) and glutathion peroxidase (metaphosphoric acid SIGMA ALDRICH y EnzyChromTM GSH/GSSG Assay Kit, measured with various commercial kits, in U/μL
Changes in lymphocyte subpopulations from baseline to 12 and 24 weeks | Baseline, 12 and 24 weeks
  Cluster of desgination 4, 8, 17 and 19 (CD4+, CD8+, CD17+ and CD19+), measured by flow cytometry (Becton Dickinson Facs AriaMR de 6 canales), in percentage
Changes in Intestinal microbiota patterns from baseline to 12 and 24 weeks | Baseline, 12 and 24 weeks
  Analyzed with a Illumina sequencing equipment and Mothur y Stamp softwares, in percentage

OTHER OUTCOMES:
Change in plasma vitamin C from baseline to 12 and 24 weeks | Baseline, 12 and 24 weeks
  Measured with a Colorimetric assay, in mg/dL
Changes in plasma vitamin D from baseline to 12 and 24 weeks | Baseline, 12 and 24 weeks
  Measured with a commercial ELISA kit, ng/mL
Changes in plasma zinc from baseline to 12 and 24 weeks | Baseline, 12 and 24 weeks
  Measured with a Colorimetric assay, in mg/dL

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Baothman+OA%2C+Zamzami+MA%2C+Taher+I%2C+ABugaker+J%2C+Abu-Farhca+MA.+The+role+of+Gut+Microbiota+in+the+development+of+obesity+and+diabetes
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Barengolts+E.+Vitamin+D+and+prebiotics+may+benefit+the+intestinal+microbacteria+and+improve+glucose+homeostasis+in+prediabetes+and+type+2+diabetes.
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Capdor+J%2C+Foster+M%2C+Petocz+P%2C+Samman+S.+Zinc+and+glycemic+control%3A+a+meta-analysis+of+randomised+placebo+controlled+supplementation+trials+in+humans.
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Fruit+and+vegetable+intake+and+the+association+with+glucose+parameters%3A+a+cross-sectional+analysis+of+the+Let%27s+Prevent+Diabetes+Study
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/15008827
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Foster+M%2C+Petocz+P%2C+Samman+S.+Inflammation+markers+predict+zinc+transporter+gene+expression+in+women+with+type+2+diabetes+mellitus
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Gokhale+NH%2C+Acharya+AB%2C+Patil+VS%2C+Trivedi+DJ%2C+Thakur+SL.+(2013)+A+short-term+evaluation+of+the+relationship+between+plasma+ascorbic+acid+levels+and+periodontal+disease+in+systemically+healthy+and+type+2+diabetes+mellitus+subjects
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Jansen+J%2C+Rosenkranz+E%2C+Overbeck+S%2C+Warmuth+S%2C+Mocchegiani+E%2C+Giacconi+R%2C+Weiskirchen+R%2C+Karges+W%2C+Rink+L.+Disturbed+zinc+homeostasis+in+diabetic+patients+by+in+vitro+and+in+vivo+analysis+of+insulinomimetic+activity+of+zinc
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/20606205
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/22699609
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Kayaniyil+S%2C+Vieth+R%2C+Retnakaran+R%2C+Knight+JA%2C+Qi+Y%2C+Gerstein+HC%2C+et+al.+Association+of+vitamin+D+with+insulin+resistance+and+beta-cell+dysfunction+in+subjects+at+risk+for+type+2+diabetes.+Diabetes+care
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Ley%2C+R.+E.%2C+Lozupone%2C+C.+A.%2C+Hamady%2C+M.%2C+Knight%2C+R.+%26+Gordon%2C+J.+I.+Worlds+within+worlds%3A+evolution+of+the+vertebrate+gut+microbiota
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Mandl+J%2C+Szarka+A%2C+Bángheyl.+(2009)+Vitamin+C%3A+update+on+physiology+and+pharmacology.+B+J+Pharmacol
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Efficacy+of+supplementary+vitamins+C+and+E+on+anxiety%2C+depression+and+stress+in+type+2+diabetic+patients%3A+a+randomized%2C+single-blind%2C+placebo-controlled+trial
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Effect+of+vitamin+C+supplementation+on+postprandial+oxidative+stress+and+lipid+profile+in+type+2+diabetic+patients.
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/9794114
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Rafighi%2C+Z.%2C+Shiva+A.%2C+Arab%2C+S.+and+Mohd+Yousof%2C+R.+(2013)+Association+of+dietary+vitamin+C+and+E+intake+and+antioxidant+enzymes+in+type+2+diabetes+mellitus+patients
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Zinc+as+a+potential+coadjuvant+in+therapy+for+type+2+diabetes.
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Sarmento+RA%2C+Silva+FM%2C+Sbruzzi+G%2C+Schaan+BD%2C+Almeida+JC.+Antioxidant+micronutrients+and+cardiovascular+risk+in+patients+with+diabetes%3A+a+systematic+review
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/25284151
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/27915988
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Insulino-mimetic+and+anti-diabetic+effects+of+zinc
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/28615382
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/12502486
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/22375253
- Available data/document: scientific article — http://www.ncbi.nlm.nih.gov/pubmed/?term=Iman+M+Ibrahim%2C+and+Manal+M+Alkady.+Role+of+Vitamin+D+on+glycemic+control+and+oxidative+stress+in+type+2+diabetes+mellitus

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT03734445/Prot_SAP_002.pdf
  • Informed Consent Form (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT03734445/ICF_003.pdf